CLINICAL TRIAL: NCT00864708
Title: Enhancing Function Using the RF Microstimulator Gait System Following Stroke 2008
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment period/study duration had exceeded The Alfred Mann Foundation's timeline.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: The Alfred E. Mann Foundation for Scientific Research (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3252-R; B3513R (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Stroke
Keywords: Functional Electrical Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): radio frequency-controlled (RF) Microstimulator (RFM) Gait System
  Interventions: Device: radio frequency-controlled (RF) Microstimulator (RFM) Gait System

INTERVENTIONS:
Device: radio frequency-controlled (RF) Microstimulator (RFM) Gait System — Fully Implanted FES system to assist patient with gait component practice

SUMMARY:
The purpose of the study is to investigate new Technology for recovery of ankle walking function after stroke.

DETAILED DESCRIPTION:
Background and Purpose: Conventional rehabilitation does not restore normal, upper limb function or normal gait to many stroke survivors. Functional neuromuscular stimulation (FNS) has shown promise for functional enhancement of both upper and lower limb motor control following stroke. Gains included muscle activation latencies, strength, coordination, upper limb functional tasks, gait kinematics, walking endurance, and quality of life. The purpose of the proposed work is to test the radio frequency-controlled (RF) Microstimulator (RFM) Gait System regarding system performance and subject response to treatment.

Methods: This is a feasibility study in which up to four subjects will receive the (RFM) Gait System. Up to ten RFMs will be placed for a given subject. An RFM ankle muscle system will be used to train ankle gait components. A separate RFM system will be used to train knee gait components. Subjects will be treated for 6 months, four sessions/wk. Primary outcome measures for the RFM Gait System will be: kinematic swing phase gait components and walking endurance. Secondary outcome measures will include: strength, coordination, spasticity, function, and quality of life. Data collections will occur at months 1, 3 and 6, and for follow-up times up to a year after the end of treatment. The results of the RFM ankle system have the potential to provide a new technology for ankle muscle gait components.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient endurance to participate in rehabilitation sessions.
* Medically Stable
* Age >21 years.
* Inability to perform normal ankle coordinated gait components.
* Participants should be able to walk and keep balance without physical assistance from another person

Exclusion Criteria:

* Acute or progressive cardiac, renal, respiratory, neurological disorders or malignancy.
* Lower motor neuron damage or radiculopathy
* Allergy or contraindication to anesthesia, Versed, (or comparable substitute.
* Active implantable device (e.g. pacemaker, implantable cardiac defibrillator, neurostimulator, or drug infusion device.
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, PhD MS, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dec 2008 - October 2009, recruitment by flier and by word of mouth
Groups:
- Arm 1: Gait training using radio frequency-controlled (RF) Microstimulator (RFM) Gait System
Period: Overall Study
Arm/Group | Arm 1
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was a feasibility study to test an RFM Gait System for re-training gait coordination. Number of participants was limited to sponsor timeline.
Groups:
- Arm 1: Gait training using radio frequency-controlled (RF) Microstimulator (RFM) Gait System )
Arm/Group | Arm 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Walking Endurance (6MWT)
Description: The Six Minute Walk Test (6MWT) is a measure of the distance measured in feet ambulated by the participant during six minutes. A further distance walked in 6 minutes indicates improvement on the measure.
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: feet
Groups:
- Arm 1: gait training with radio frequency-controlled (RF) Microstimulator (RFM) Gait System
Arm/Group | Arm 1
Number analyzed (Participants) | 1
feet
  Day 1-6MWT | 843
  After 3 months of treatment- 6MWT | 771

2. Secondary Outcome: Fugl-Meyer Lower Extremity Score
Description: Fugl-Meyer Lower Extremity Score (FMLE) is an itemized measure of lower extremity coordination following stroke. Scores for the FMLE range from 0 (most impaired) to 34 (normal).
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 1
units on a scale
  Day 1- Fugl Meyer Score | 22
  After 3 months of treatment- Fugl Meyer Score | 26

3. Secondary Outcome: Ashworth Scale
Description: The Ashworth Scale is a measure of muscle spasticity; muscle groups are graded from 0 (no spasticity) to 4 (greatest spasticity/contracture). The lower limb muscle groups are summed for a total lower limb Ashworth score. A lower score indicates better performance. (range is 0-40)
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 1
units on a scale
  Day 1-Ashworth Score | 1.5
  After 3 months of treatment- Ashworth Score | 1.0

4. Secondary Outcome: Stroke Impact Scale (SIS)
Description: The SIS is a measure of Quality of Life/Life Role Participation following stroke. Each item in a domain is scored between 0 and 5. A higher score indicates better performance (range 0-295).
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 1
units on a scale
  Day 1-SIS | 261
  After 3 months of treatment- SIS | 264

5. Secondary Outcome: Manual Muscle Testing (MMT)
Description: This is a measure of strength of the various muscle groups of the lower limb. Each is graded on a 0 to 5 scale; the final score is the summed total of the lower limb muscle groups tested. (score range of summed muscles is 0-50, with 50 being the maximum highest score)
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 1
units on a scale
  Day 1-MMT | 21.35
  After 3 months of treatment- MMT | 23.33

6. Primary Outcome: Kinematic Gait Measures
Description: assessment of the lower limb kinematics during ambulation at chosen speed.
Time Frame: Day 1 and at 3 months, following treatment
Measure: Number; unit: percentage of change Day 1 to 3 months
Arm/Group | Arm 1
Number analyzed (Participants) | 1
percentage of change Day 1 to 3 months | 0

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=1)
delivery of unactivated stimuli (within comfort) (Musculoskeletal and connective tissue disorders) | 1 (1) — RFM system delivered unactivated stimuli (always reported within comfort) to subject unpredictably at times when system was powered up. AMF submitted device re-test data and reports to FDA which then re-approved continued use of the RFM system.

LIMITATIONS AND CAVEATS:
Study sponsor, Alfred Mann foundation (AMF) stopped study because "enrollment period/study duration has exceeded the AMF's timeline".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are employed by the Department of Veterans Affairs (DVA) which funded the study; the Alfred P. Mann Foundation (AMF) provided the technology that was tested.

There was an agreement between the Principal Investigators of the DVA and the AMF that the AMF would be provided a period of time to review any manuscript for publication and provide input. There was no restriction regarding PI's rights to discuss or publish the results.